CLINICAL TRIAL: NCT03488667
Title: A Phase II Study of Perioperative mFOLFOX (Fluorouracil, Leucovorin, and Oxaliplatin) Chemotherapy Plus Pembrolizumab(MK-3475) Combination in Patients With Potentially Resectable Adenocarcinoma of the Gastroesophageal Junction (GEJ) and Stomach (MISP #52216)
Brief Title: Perioperative mFOLFOX Plus Pembrolizumab in Gastroesophageal Junction (GEJ) and Stomach Adenocarcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-2017-PeriopmFOLFOXPem
Record Dates: First submitted 2018-03-28; First posted 2018-04-05 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Gastro Esophageal Junction Cancer; Stomach Cancer; Adenocarcinoma
Keywords: resectable adenocarcinoma of Gastroesophageal Junction; resectable adenocarcinoma of Stomach
MeSH Terms: conditions — Stomach Neoplasms; Adenocarcinoma | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- mFOLFOX6 (Leucovorin-Fluorouracil-Oxaliplatin) + Pembrolizumab (Experimental): Drug: Pembrolizumab Dose: 200 mg Dose Frequency: Every three weeks (Q3W) Route: Intravenous (IV) infusion
  Drug: Oxaliplatin Dose: 85 milligrams per meter squared (mg/m2) Dose Frequency: Every 2 weeks (Q2W) Route: IV infusion
  Drug: Leucovorin Dose: 400 mg/m2 Dose Frequency: Q2W Route: IV infusion
  Drug: Fluorouracil Dose: 400 mg/m2 Dose Frequency: Q2W Route: IV bolus
  Drug: Fluorouracil Dose: 2,400 mg/m2 Dose Frequency: Q2W Route: IV continuous 46-hour infusion
  Pembrolizumab will be administered at a fixed dose of 200 mg IV over 30 minutes every 3 weeks. Participants will receive 3 doses of the drug on Days 1, 22, 43 during the neoadjuvant phase of the study, and 12 doses of the drug on Days 1, 22, 43 during the adjuvant phase of the study (total 15 doses). Participants will receive 4 doses of mFOLFOX6 regimen on Days 1, 15, 29, 43 during the neoadjuvant phase of the study, and 4 doses during the adjuvant phase of the study (total 8 doses).
  Interventions: Drug: Neoadjuvant Treatment - mFOLFOX6 & Pembrolizumab; Drug: Adjuvant Treatment - mFOLFOX & Pembrolizumab

INTERVENTIONS:
Drug: Neoadjuvant Treatment - mFOLFOX6 & Pembrolizumab — Pembrolizumab, mFOLFOX Chemotherapy
Drug: Adjuvant Treatment - mFOLFOX & Pembrolizumab — Pembrolizumab, mFOLFOX Chemotherapy

SUMMARY:
To evaluate the antitumor activity and safety/tolerability of the combination (mFOLFOX + Pembrolizumab) in patients with potentially resectable adenocarcinoma of the Gastroesophageal Junction (GEJ) and stomach.

DETAILED DESCRIPTION:
This study will evaluate the efficacy and safety of perioperative mFOLFOX plus Pembrolizumab combination regimen in participants with potentially resectable adenocarcinoma of the GEJ and stomach.

* The study is a non-randomized, open-label, single-arm phase II study.
* The enrolled participants will receive neoadjuvant combination of mFOLFOX every 2 weeks for 4 doses (on Days 1, 15, 29, 43) and Pembrolizumab every 3 weeks for 3 doses (on Days 1, 22, 43).
* Serious adverse events (SAEs) will be assessed on an ongoing basis using CTCAE v4.0, and the Thall, Simon, and Estey's design to monitor the efficacy and toxicity continuously together.
* Repeat PET-CT will be obtained approximately 2-3 weeks after completion of neoadjuvant combination therapy.
* If no evidence of metastatic disease on PET-CT, participants will undergo potentially curative surgical resection 4-6 weeks after completion of neoadjuvant combination therapy. This will be followed by adjuvant combination therapy (to be started 6-8 weeks after surgery) consisting of mFOLFOX every 2 weeks for additional 4 doses (total 4 months of therapy) plus Pembrolizumab every 3 weeks for additional 12 doses (total 1 year of therapy). If there is evidence of metastatic disease on PET-CT, participant will come off the study (i.e., will not undergo surgical resection and adjuvant therapy).
* Participants will continue to receive treatment until either one of the following occurs: completion of adjuvant therapy, development of radiographically confirmed progression, participant withdraws consent, intercurrent illness that prevents further administration of treatment, or sponsor-investigator decides to withdraw the participant.
* Efficacy outcomes during the adjuvant chemotherapy phase will be determined by radiologic measurements by CT using RECIST v1.1. Assessment of response will be performed every 3 months for the first year and as per the standard institutional guidelines thereafter.

ELIGIBILITY:
Inclusion Criteria:

1. Male/female participants who are 18 - 75 years of age on the day of signing informed consent with histologically or cytologically confirmed diagnosis of adenocarcinoma of the gastroesophegeal junction (GEJ) or stomach will be enrolled in this study.
2. Have newly diagnosed localized or locally advanced, potentially resectable disease without any prior systemic chemotherapy.
3. Have no evidence of distant metastases.
4. Be eligible and reasonably fit to undergo potentially curative resection

   Male participants:
5. A male participant must agree to use a contraception as detailed in Appendix 3 of this protocol during the treatment period and for at least 120 days after the last dose of study treatment and refrain from donating sperm during this period. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the participant.

   Female participants:
6. Female participants of childbearing potential must have a negative serum pregnancy within 72 hours prior to enrollment.
7. A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

   1. Not a woman of childbearing potential (WOCBP) OR
   2. A WOCBP who agrees to follow the contraceptive guidance in Appendix 3 during the treatment period and for at 120 days after the last dose of study treatment. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the participant.
8. The participant (or legally authorized representative, if applicable) must be willing and able to provide written informed consent for the trial.
9. Have evaluable disease . Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
10. Have pre-resection tissue available.
11. Be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion.
12. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
13. Have adequate organ function.
14. Be willing to provide blood and tissue samples for research purposes.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

1. A WOCBP who has a positive serum pregnancy test within 72 hours prior to enrollment on study.
2. Has received prior therapy with an anti-PD-1 (Programmed death-1), anti-PD-L1 (programmed death ligand-1), or anti PD L2 (programmed death ligand-2) agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor.
3. Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks prior to study enrollment.
4. Has received prior chemotherapy (including investigational agents) for any malignant disorder, thoracic radiation therapy or prior surgical resection of an esophagogastric tumor.

   a. Note: If participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment.
5. Has received prior radiotherapy within 2 weeks of start of study treatment. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis.
6. Has biopsy-proven invasion of tracheobronchial tree or tracheo-esophageal fistula.
7. Has distant metastatic disease on imaging or staging laparoscopy at the time of study entry.
8. Has a known history of active TB (tuberculosis)
9. Hypersensitivity to pembrolizumab or any of its excipients.
10. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered from adverse events due to agents administered more than 4 weeks earlier.
11. Clinically significant peripheral neuropathy at the time of study entry.
12. Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines are live attenuated vaccines and are not allowed.
13. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.

    a. Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.
14. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
15. Has a known additional malignancy that is progressing or has required active treatment within the past 3 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g. breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
16. Has active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically serious autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment. Participants with vitiligo or resolved childhood asthma/atopy would be an exception to this rule. Participants that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Participants with hypothyroidism stable on hormone replacement or Sjogren's syndrome will not be excluded from the study.
17. Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
18. Has an active infection requiring systemic therapy.
19. Has a known history of Human Immunodeficiency Virus (HIV).
20. Has a known history of Hepatitis B or known active Hepatitis C virus infection. Note: testing for Hepatitis B and Hepatitis C is required only if mandated by local health authority.
21. Inoperable on the basis of co-existent medical problems.
22. Non-malignant systemic disease (cardiovascular, renal, hepatic, etc.) that would preclude any of the study drugs.
23. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator.
24. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
25. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-06-27 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Pathological response rate (ypRR) | 10-14 weeks
  Number of participants with ypRR after neoadjuvant therapy. Will be assessed on the surgical resection specimen after neoadjuvant therapy, using Haemotoxylin and Eosin (H&E) staining and evaluated using Tumor Regression Score.
Number of Adverse Events related to toxicity. | up to 14 months
  Number of participants with adverse events related to toxicity. Evaluated using Common Terminology Criteria for Adverse Events (CTCAE) version 4.03. Participants will be followed for adverse event monitoring through the final safety follow up visit or until study discontinuation/disease progression, whichever occurs first.

SECONDARY OUTCOMES:
Objective response rate (ORR) | 12 months
  Number of participants with ORR (partial response and complete response) at 12 months. Evaluated using RECIST v1.1
Disease Free Survivial (DFS) | 12 months
  Number of participants with DFS. Evaluated using computed tomography (CT).
Overall Survival (OS) | 12 months
  Number of participants with OS.
PET response rate after completion of neo-adjuvant therapy. | 10 weeks
  Evaluated using Positron emission tomography scan & computed tomography (PET-CT)
Programmed cell death ligand 1 (PD-L1) expression in tumor cells | baseline and between 16-21 weeks
  Change in PD-L1 expression on the surface and in the nucleus of the tumor cells over treatment will be related to complete pathological response (ypCR) by means of logistic regression. Evaluated by immunohistochemistry (IHC). Participants will be evaluated at baseline and reevaluated 2-4 weeks after surgery (for those participants who develop complications from surgery, the revaluation time frame may be extended to 7 weeks).

CONTACTS AND LOCATIONS:
Overall Officials: Weijing Sun, MD, FACP, Principal Investigator — The University of Kansas - Cancer Center
Locations (1):
- The University of Kansas Cancer Center, Westwood, Kansas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chang X, Ge X, Zhang Y, Xue X. The current management and biomarkers of immunotherapy in advanced gastric cancer. Medicine (Baltimore). 2022 May 27;101(21):e29304. doi: 10.1097/MD.0000000000029304. PMID 35623069